CLINICAL TRIAL: NCT01345201
Title: A Phase 1 Dose Escalation Study of OMP-18R5 in Subjects With Solid Tumors
Brief Title: A Dose Escalation Study of OMP-18R5 in Subjects With Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: OncoMed Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Organization: Mereo BioPharma (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 18R5-001
Record Dates: First submitted 2011-04-27; First posted 2011-04-29 (Estimated); Last update posted 2020-09-09 (Actual); Status verified 2020-09

CONDITIONS: Solid Tumors
Keywords: Phase 1; dose escalation; histologically confirmed; malignancy metastatic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Biological: OMP-18R5 — IV infusion. Subjects with stable disease or a response at Day 56 will be allowed to continue until disease progression.

SUMMARY:
This is an open-label Phase 1 dose escalation study of OMP-18R5 in subjects with a solid tumor for which there is no remaining standard curative therapy and no therapy with a demonstrated survival benefit. Up to 44 subjects will be enrolled at up to 2 centers. Subjects will be assessed for safety, immunogenicity, pharmacokinetics, biomarkers, and efficacy. No formal interim analyses will be performed.

Prior to enrollment, subjects will undergo screening to determine study eligibility. Upon enrollment, subjects will receive intravenous (IV) infusions of OMP-18R5 at a assigned dosing schedule for 56 days. After 56 days, subjects will be assessed for disease status. If there is no evidence of disease progression or if the tumor is smaller, then subjects may continue to receive IV infusions of OMP-18R5 every week until disease progression.

Dose escalation will be conducted to determine the maximum tolerated dose (MTD). No dose escalation or reduction will be allowed within a dose cohort. The first 2 subjects enrolled in a cohort will not be treated on the same day. The dose may be administered at any time during the day. Three subjects will be treated at each dose level if no dose-limiting toxicities (DLTs) are observed. If 1 of 3 subjects experiences a DLT, that dose level will be expanded to 6 subjects. If 2 or more subjects experience a DLT, no further subjects will be dosed at that level and 3 additional subjects will be added to the preceding dose cohort unless 6 subjects have already been treated at that dose level. Subjects will be assessed for DLTs from the time of the first dose through 28 days. Dose escalation for newly enrolled subjects, if appropriate, will occur after all subjects in a cohort have completed their Day 28 DLT assessment. Subjects with stable disease or a response at Day 56 will be allowed to continue to receive weekly doses of OMP-18R5 until disease progression. An additional 14 subjects will be enrolled at the highest dose level that result in < 2 of the 6 subjects experiencing a Grade 3 (not including a Grade 3 infusion reaction that resolves in 24 hours) or 4 adverse event (DLT).

ELIGIBILITY:
Inclusion Criteria:

1. Subjects must have a histologically confirmed malignancy that is metastatic or unresectable for which there is no remaining standard curative therapy and no therapy with a demonstrated survival benefit. In addition, subjects must have a tumor that is at least 1 cm in a single dimension and is radiographically apparent on CT or MRI.
2. Subjects must have received their last chemotherapy, biologic, or investigational therapy at least 4 weeks prior to enrollment, 6 weeks if the last regimen included BCNU or mitomycin C.
3. Age >18 years
4. ECOG performance status <2 (see Appendix B)
5. Life expectancy of more than 3 months
6. Subjects must have adequate organ and marrow function as defined below:

   Absolute neutrophil count >1000/µL Hemoglobin >9.0 g/dL Platelets >100,000/µL Total bilirubin <1.5 X institutional upper limit of normal (ULN) AST (SGOT) and ALT (SGPT) < 3 X institutional ULN (for subjects with hepatic metastases < 5 X institutional ULN) PT and PTT within 1.5 X institutional ULN Creatinine <1.5 X institutional ULN OR Creatinine clearance >60 mL/min/1.73 m2 for subjects with creatinine levels above institutional normal
7. Women of childbearing potential must have had a prior hysterectomy or have a negative serum pregnancy test and be using adequate contraception prior to study entry and must agree to use adequate contraception from study entry through at least 6 months after discontinuation of study drug. Men must also agree to use adequate contraception (barrier method of birth control, abstinence) prior to study entry and from study entry through at least 6 months after discontinuation of study drug. Should a woman enrolled in the study or a female partner of a man enrolled in the study become pregnant or suspect she is pregnant while participating in this study or within 6 months after discontinuation of study, she should inform the Investigator immediately.
8. Ability to understand and the willingness to sign a written informed consent document

Exclusion Criteria:

1. Subjects receiving any other investigational agents
2. Subjects with brain metastases (subjects must have a CT scan or MRI of the head within 28 days prior to enrollment to rule out brain metastases), uncontrolled seizure disorder, or active neurologic disease
3. History of a significant allergic reaction attributed to humanized or human monoclonal antibody therapy
4. Significant intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements
5. Pregnant women or nursing women
6. Subjects with known HIV infection
7. Known bleeding disorder or coagulopathy
8. Subjects receiving heparin, warfarin, or other similar anticoagulants, except for subjects on low molecular weight heparin for DVT/PE prophylaxis. Note: Subjects may be receiving low-dose aspirin and/or non-steroidal anti-inflammatory agents.
9. New York Heart Association Classification III, or IV (see Appendix D)
10. Subjects with known clinically significant gastrointestinal disease including, but not limited to, inflammatory bowel disease.
11. Subjects with known osteopenia or osteoporosis.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2011-05; Primary Completion 2014-05 (Actual); Study Completion 2014-05 (Actual)

PRIMARY OUTCOMES:
To determine the safety of OMP-18R5 in subjects with previously treated solid tumors | Subjects will be assessed for dose limiting toxicity from Days 0-28. Adverse events will be reported through 30 days after the last dose.

SECONDARY OUTCOMES:
To determine the pharmacokinetics of OMP-18R5 in subjects with previously treated solid tumors | The first 8 weekly doses and following treatment termination
  The half-life, volume of distribution, and clearance will be determined.
To determine the immunogenicity of OMP-18R5 in subjects with previously treated solid tumors | Subjects will be assessed during screening, every 4 weeks, treatment termination, weekly for the first 4 weeks following d/c of study drug, Weeks 8 and 12 following d/c of drug.
To assess the preliminary efficacy of OMP-18R5 in subjects with previously treated solid tumors | Every 56 days until disease progression
  The response outcome in patients will be determined.

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - UCLA Santa Monica Hematology-Oncology, Santa Monica, California
  - University of Michigan Health System, Ann Arbor, Michigan
  - South Texas Accelerated Research Therapeutics, San Antonio, Texas